CLINICAL TRIAL: NCT07110454
Title: A Prospective Long-Term Follow-Up Study to Evaluate the Use of the Minder Device to Aid in Treatment After Actionable Event Identification in Patients Diagnosed With Epilepsy.
Brief Title: Diagnosing Epilepsy To EffeCT Change Long-Term Follow-Up
Acronym: DETECT LTFU
Status: Recruiting | Type: Observational
Sponsor: Epiminder America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EM2402
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Epilepsy (Treatment Refractory)
Keywords: Minder System; Sub-scalp EEG monitoring device
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational: Minder System
  Interventions: Device: Previous receipt of the Minder System (implantable continuous electroencephalographic (EEG) monitoring (iCEM) system)

INTERVENTIONS:
Device: Previous receipt of the Minder System (implantable continuous electroencephalographic (EEG) monitoring (iCEM) system) — The Minder System consists of an implanted device containing an electrode lead and telemetry unit. The electrode lead contains four electrodes that are placed under the patient's scalp to record electrical activity (EEGs) from both sides of the brain. The electrode lead is connected to the telemetry until that continuously transmits these signals to the external Minder devices to remotely show EEGs for clinician review.

SUMMARY:
The purpose of this research is to address the challenges of correctly monitoring, managing, and diagnosing epilepsy in participants whose seizures are not well captured by standard electroencephalography (EEG) tests and who cannot use or are not able to use more standard monitoring techniques. This research is being done to understand how the Minder System helps physicians make decisions about participant's epilepsy treatment after an actionable event. The Minder System was granted De Novo classification by the U.S. Food and Drug Administration (FDA) and is not investigational.

Participants that have completed the DETECT study and received the Minder System previously will consent to join this long-term follow-up observational study. The study will collect information about general wellbeing, use of healthcare services, and experience using the Minder data over time to support long-term epilepsy care.

All participants will continue to be followed by their treating physician and undergo assessments and visits every six (6) months until two (2) years after receiving the Minder device.

ELIGIBILITY:
Inclusion Criteria:

* Participant met all inclusion criteria, was enrolled in the DETECT study, and received the Minder device
* Participant completed the DETECT study by receiving an actionable event or by completing the 6-month follow-up visit
* Participant continues to have the Minder device implanted
* Participant must continue to meet relevant DETECT study inclusion criteria

Exclusion Criteria:

* Participant meets any relevant DETECT study exclusion criteria including needing treatments or assessments that are not indicated with the Minder System like Magnetic Resonance Imaging (MRI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants previously implanted with the Minder device
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Minder System to aid in treatment following an actionable event by comparing change using the Patient Global Impression scale (PGIC) from baseline to follow-up. | 2 years

OTHER OUTCOMES:
To evaluate the Minder System to aid in treatment following an actionable event by comparing change using Clinician Global Impression scale (CGIC) from baseline to follow-up. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing quality of life using the EQ-5D from baseline to follow-up. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing healthcare utilization by number of surgeries or procedures. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing healthcare utilization by medication usage. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing healthcare utilization by the number of hospital visits. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing participant wellbeing using the Beck Anxiety Inventory (BAI) for symptoms associated with anxiety from baseline to follow-up. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing participant wellbeing using the Beck Depression Inventory (BDI) for symptoms associated with depression from baseline to follow-up. | 2 years
To evaluate the Minder System to aid in treatment following an actionable event by comparing quality of life using the Quality of life in epilepsy-31 (QOLIE-31) from baseline to follow-up. | 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halliday AJ, Gillinder L, Lai A, Seneviratne U, Fontenot H, Cameron T, McLean K, Niemiec A, Raghupathi R, Ganguly TM, Ellis C, Conrad EC, Briggs R, Bulluss K, Kwan P, Perucca P, O'Brien TJ, McGonigal A, Gutman M, Papacostas J, Fong MWK, Lee A, Crompton DE, Laing J, Wijayath M, Morokoff AP, Murphy M, D'Souza WJ, Cook MJ. The UMPIRE study: A first-in-human multicenter trial of bilateral subscalp monitoring for epileptic seizure detection. Epilepsia. 2025 Sep;66(9):3426-3439. doi: 10.1111/epi.18458. Epub 2025 May 30. PMID 40445205